CLINICAL TRIAL: NCT01463865
Title: Selective Block of the Axillary Nerve in Postoperative Pain Management, a Randomised, Blinded, Placebo-controlled Trial
Brief Title: Selective Block of the Axillary Nerve in Postoperative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Kai Henrik Wiborg Lange, Head of research, Associate professor, phd, Hillerod Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1-2011-057
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Sodium chloride
  Interventions: Drug: Sodium chloride
- ropivacaine (Active Comparator): Naropin
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — Single shot nerve block with ropivacaine 10-20 ml; 7,5 mg/ml
  Other Names: Naropin
  Arms: ropivacaine
Drug: Sodium chloride — Single shot nerve block with isotonic sodiumchloride 10-20 ml; 0.9%
  Arms: Placebo

SUMMARY:
In this study the investigators wish to compare the effect of a selective axillary nerve block to placebo in patients undergoing arthroscopic shoulder surgery.

It is the investigators hypothesis that the amount of morphine consumption in the first 4 hours postoperatively in the intervention group will be significant lower than in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing arthroscopic shoulder surgery
* Age between 18 and 80 years
* ASA 1-3
* BMI between 18 and 35 kg/m2
* Subjects which have given their written informed consent

Exclusion Criteria:

* Subjects unable to cooperate to the investigation
* Subjects not understanding or speaking danish
* Subjects allergic to intervention drugs
* Daily use of strong analgesics (morphine, oxycontine, ketogan)
* Alcohol or medicine misuse
* Failure of nerve block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 0-4 hours postoperatively
  Patients are coupled to an intravenous PCA pump. The amount of morphine administered by the patient in the first 4 hours postoperatively is registered.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) score | 0-12 hours and 12-24 hours postoperatively
  Postoperative VAS scores during the first 24 hours postoperatively, divided into two periods.
Total morphine consumption | 0-24 hours postoperatively
  The total amount of morphine administered during the first 24 hours postoperatively
Postoperative nausea and vomiting (PONV) | 0-4, 0-12 and 12-24 hours postoperatively
  Postoperative nausea evaluated on a 1-3 scale with and without vomiting
Escape block | 0-4 hours postoperatively
  The use of an escape block (interscalene brachial plexus block) in patients with pain breakthrough despite IV morphine 0-4 hours postoperatively.
Bolus morphine 5 mg iv | 0-4 hours postoperatively
  Number of morphine boli administered during the first 4 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Aleris-Hamlet Hospital, Frederiksberg, Denmark

REFERENCES:
- [Background] Rothe C, Asghar S, Andersen HL, Christensen JK, Lange KH. Ultrasound-guided block of the axillary nerve: a volunteer study of a new method. Acta Anaesthesiol Scand. 2011 May;55(5):565-70. doi: 10.1111/j.1399-6576.2011.02420.x. PMID 21827442
- [Derived] Rothe C, Lund J, Jenstrup MT, Steen-Hansen C, Lundstrom LH, Andreasen AM, Lange KHW. A randomized controlled trial evaluating the impact of selective axillary nerve block after arthroscopic subacromial decompression. BMC Anesthesiol. 2020 Jan 31;20(1):33. doi: 10.1186/s12871-020-0952-y. PMID 32005160